CLINICAL TRIAL: NCT04636411
Title: Evaluation of the Effects of Oral Magnesium Supplementation on Glycemic Control and Inflammation Among Patients With Type 2 Diabetes
Brief Title: Effects of Oral Magnesium Supplementation on Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samar Fares, MD (Other)
Collaborators: Walaa Reda Abdel Fattah Mohamed Badr (Unknown); Marwa Mostafa Ahmed (Unknown); Moushira Hosny Ezzelarab Sayed (Unknown); Nagwa Eid Sobhy Saad (Unknown)
Responsible Party: Sponsor-Investigator, Samar Fares, MD, Lecturer of family medicine, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-164-2020
Record Dates: First submitted 2020-11-08; First posted 2020-11-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Type2 Diabetes
Keywords: Oral Magnesium; Type 2 Diabetes; Diabetes Control; HbA1c; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study participants will be randomized into 2 groups (intervention and control group) to be studied simultaneously
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group group will receive oral magnesium supplementation (250 mg of elemental magnesium daily for three months) plus the standard care for diabetic patients
  Interventions: Dietary Supplement: Oral Magnesium Supplementation; Other: Standard Care for diabetic patients
- Control group (Active Comparator): This group will receive the standard care for diabetic patients
  Interventions: Other: Standard Care for diabetic patients

INTERVENTIONS:
Dietary Supplement: Oral Magnesium Supplementation — 250 mg of elemental magnesium daily for three months
  Arms: Intervention group
Other: Standard Care for diabetic patients — Health education, oral antihyperglycemic medications according to American Diabetes Association (ADA) guidelines

SUMMARY:
A total of 74 Adult Patients with type 2 diabetes mellitus (T2D) will be enrolled and randomized into 2 groups. The intervention group will receive oral magnesium (Mg) supplementation. The study objectives are:

1. To estimate level of Mg (total and ionized) in patient with type 2 DM.
2. To determine the effect of Mg supplementation for diabetic patient on serum Mg level, glycemic control and level of inflammation.
3. To assess the correlation between serum Mg level and glycemic control and level of inflammatory mediators (CRP)

DETAILED DESCRIPTION:
A total of 74 Adult Patients of both genders who had been diagnosed with T2D and are on oral anti-hyperglycemic drug and their HbA1C between 7and 8 %, will be enrolled in the study. Initially the study protocol will be explained & informed written consent will be obtained from all participants. All subjects will be evaluated to ensure that they meet the eligibility criteria through: Full history taking, complete physical examination and investigations. the intervention group will receive oral magnesium (Mg) supplementation for 3 months (250 mg of elemental magnesium daily). The primary outcome is to determine the effect of Mg supplementation for diabetic patient on serum Mg level, glycemic control and level of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes with HbA1C between 7 and 8%.
* Both genders will be included in this study.

Exclusion Criteria:

* Patients on insulin.

  * Patients on diuretics or angiotensin-converting enzyme inhibitors in the last 2 weeks.
  * Patients taking Mg containing supplements within 3 months.
  * Patients with significant gastrointestinal disorders (eg, chronic diarrhea).
  * Patients with impaired renal functions (eGFR< 60 mL/min).
  * Heart block or heart failure
  * Patients treated with aldosterone antagonists.
  * Pregnant patients
  * Patients with evidence of infection.
  * Patients with chronic inflammatory conditions eg, SLE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 3 months
  To determine the effect of oral Mg supplementation for diabetic patient on Glycemic control
Inflammation | 3 months
  To determine the effect of oral Mg supplementation for diabetic patient on inflammation (CRP)

SECONDARY OUTCOMES:
Serum magnesium level | 3 months
  To determine the effect of Mg supplementation for diabetic patient on serum Mg level
Prevalence of hypomagnesemia | up to 4 weeks
  To estimate prevalence of hypomagnesemia in patients with type 2 DM.
Correlation of serum Mg level | up to 4 weeks
  To assess the correlation between serum Mg level and glycemic control and level of inflammatory mediators (CRP).
Total or ionized Mg | 3 months
  Determine the more accurate measure for Mg in diabetic patient either total or ionized Mg

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa E Saad, Professor, Principal Investigator — Cairo University
Locations (1):
- Mokattam primary health care unit, Cairo, Mokattam, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study data will be available upon reasonable request from central contact person
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After finalizing the study
Access Criteria: The study data will be available upon reasonable request from central contact person

REFERENCES:
- [Background] Saeed H, Haj S, Qasim B. Estimation of magnesium level in type 2 diabetes mellitus and its correlation with HbA1c level. Endocrinol Diabetes Metab. 2018 Nov 2;2(1):e00048. doi: 10.1002/edm2.48. eCollection 2019 Jan. PMID 30815575
- [Background] Dhawan S, Natarajan R. Epigenetics and Type 2 Diabetes Risk. Curr Diab Rep. 2019 Jun 27;19(8):47. doi: 10.1007/s11892-019-1168-8. PMID 31250127
- See also: Estimation of magnesium level in type 2 diabetes mellitus and its correlation with HbA1c level — http://pubmed.ncbi.nlm.nih.gov/30815575/
- See also: Epigenetics and Type 2 Diabetes Risk — http://pubmed.ncbi.nlm.nih.gov/31250127/